CLINICAL TRIAL: NCT04247711
Title: On Track Chile For First Episode Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Universidad de O'Higgins (Other); Columbia University (Other); Washington University School of Medicine (Other); New York University (Other); Research Foundation for Mental Hygiene, Inc. (Other); New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Rubén Alvarado, Associate Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH115502-02 (NIH)
Record Dates: First submitted 2020-01-10; First posted 2020-01-30 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Psychosis
Keywords: First-Episode Psychosis; Implementation Science; Coordinated Specialty Care; Global Mental Health
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The 21 participating clinics will be divided into two groups based on poverty level of catchment area and expected enrollment of individuals with FEP for each clinic. The largest site will be matched with two clinics of similar poverty level and clinic size. The matching will be done based on visual inspection of a scatter plot of expected enrollment by income of each site. The nearest neighbor matching approach will be used to choose pairs. Blocks of size 2, and one block of size 3, will be randomly generated. This procedure will entail 1) generating a random number 0 or 1 ten times, and 2) assigning 0 to the Usual FEP care clinic and 1 to the OTCH clinic in each matched pair. For the block of size 3, two sites will be assigned to either OTCH or Usual FEP care, and the remaining site to either OTCH or Usual FEP care as well. The random allocation will enable us to bring into the study one OTCH and one Usual FEP Care clinic per month (except for the block of size 3, as noted above).
Who Masked: Outcomes Assessor
Masking Description: A two-fold strategy will be used to keep the blind. First, external interviewers with experience in conducting clinical evaluations will be hired and trained. These interviewers will be blind to study hypotheses and participant assignment. A mental health professional at each clinic (ie., "Local Coordinator") will do the consent procedures and a member of the Research Staff (ie., "Registration Designee") will randomly assign consented participants to the interviewers. The latter will be blinded to treatment allocation. Second, every assessment will be conducted at a location different from the clinic where a participant receives treatment. This location could be the participant's home, an office in UOH or UCH, or any place in the community where the participant feels comfortable (e.g., a park). This approach was successfully used in a previous U-19 study led by this research team in which most of the follow-up assessments were conducted in participants' neighborhoods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTCH (Experimental): OTCH is based on OTNY, a Coordinated Specialty Care program for people with first-episode psychosis. The program is implemented by a multidisciplinary team, who provide coordinated, evidence-based services based on the interests, needs, and preferences of each participant.
  Interventions: Behavioral: OTCH
- Usual FEP services (Placebo Comparator): This is generally provided in mental health outpatient clinics which serve a population enrolled in the public health care system.
  Interventions: Behavioral: Usual FEP Services

INTERVENTIONS:
Behavioral: OTCH — OTCH is structured in three phrases (i. engagement and initial needs assessment, ii. ongoing intervention and monitoring, and iii. transition to long-term services) and lasts an average of two years. OTCH will maintain the central characteristics of the OnTrack model, as well as its core principles, which include (1) Person-centered care, (2) Shared decision-making, (3) Recovery orientation, and (4) Culturally-competent care.
  Arms: OTCH
Behavioral: Usual FEP Services — These include services such as psychiatric medication, psychotherapy, and psychoeducation for people with FEP and are usually provided at outpatient mental health clinics.
  Arms: Usual FEP services

SUMMARY:
Substantial data support early interventions for people experiencing First Episode Psychosis (FEP) to ameliorate symptoms and minimize disability. FEP programs have been widely and successfully implemented in high-income countries. With the partial exception of Chile, however, there is not a single low-and-middle-income country (LMIC) that offers universal access to FEP services. Chile is unique among LMICs in having created a platform for the implementation of FEP services, including 1) an FEP policy that mandates identification of FEP individuals at primary care and delivery of community-based FEP treatments at outpatient mental health clinics, and 2) a public health care system within which this mandate can be fulfilled. Nonetheless, previous research has documented that FEP services provided at mental health clinics do not conform to recently established evidence-based approaches. Therefore, the overarching goal of this proposal is to address the shortfall in evidence-based practices for FEP in Chile by first adapting OnTrackChile (OTCH) from OnTrackNY (OTNY), a coordinated specialty care program for FEP currently being implemented across the US, and then implementing OTCH on a wide scale. Like most FEP programs, OTNY is clinically effective, but unlike most others, it also has a well-established training and technical assistance infrastructure, and a proven track record of being scaled up in large urban areas. To achieve this goal, the Dynamic Adaptation Process will be used to first inform the adaptation and implementation of OTCH in the Chilean context. Then, a Hybrid Trial design will be employed to evaluate the implementation of OTCH as well as its effectiveness and cost in a cluster-randomized controlled trial (RCT) (N = 300 from 21 outpatient clinics). The OnTrackChile program will be offered in half of these outpatient clinics; usual care services will continue to be offered at the other clinics. Study participants (ages 15 to 35) attending an outpatient clinic assigned to the intervention arm will receive the OTCH coordinated services provided by an interdisciplinary team, based on the interests, needs, and preferences of each study participant. Study participants attending outpatient clinics assigned to "usual care" will receive the usual services offered to people with a wide range of mental health conditions, not just those experiencing first-episode psychosis. The study will engage participants over the course of two years, with interviews to evaluate their experiences at the beginning of their participation, and again after 12 months and 24 months. Over the course of the study, 4-5 mental health providers will also be interviewed at each of the participating clinics (up to 105 additional interviews at the three timepoints). The data collected in this study will help researchers evaluate the effectiveness and cost of FEP treatments based in outpatient clinics and factors which may help or hinder these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have FEP (First Episode Psychosis)
* Individuals who are receiving services at a participating outpatient mental health clinic.
* Individuals who meet ICT-10 criteria for a diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, delusional disorder, brief psychotic disorder, or psychosis not otherwise specified.
* Individuals who have the capacity to provide fully informed consent. (For those under age 18, capacity to provide assent plus informed consent of parent/guardian.)
* Individuals who are able to participate in research assessments in Spanish

Exclusion Criteria:

* Individuals who have a non-psychiatric medical condition that impairs functioning.
* Individuals who have a psychosis due solely to another medical condition.
* Individuals who have a psychosis due to a developmental disability.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Adapted version of the OTNY Fidelity Scale | 24 months
  This scale will assess the degree to which the participating clinics deliver OTCH. The scale 24 dimensions rated on a 3-score rating where 0=unmet, 1=partially met, and 2=totally met. Higher scores mean better Fidelity.
Change on Providers' attitudes using the Evidence-Based Practice Attitude Scale | baseline, 12 months, 24 months
  Providers' attitudes to evidence-based practices will be measured by the evidence-based attitude scale (EBPAS). The EBPAS consists of 15 items rated on a five-point scale from 0=Not at all to 4=Very great extent. Higher scores mean better attitudes to evidence-based practices.
Change on Adoption of OTCH among patients using the CollaboRATE | baseline, 12 months, 24 months
  This is a 3-item scale rated on a ten-point scale from 0=No effort was made to 9=Every effort was made. Higher scores mean better Adoption.
Change on Adoption of OTCH among providers using the Shared Decision Making Questionnaire Physician Version | baseline, 12 months, 24 months
  This questionnaire continues with nine items about the steps in the adoption of the shared-decision making approach, one of the key components of OTCH. Each item is rated on a six-point scale from 0=Completely disagree to 5=Completely agree. Higher scores indicate more shared-decision making.
Change on Adoption of OTCH among both patients and providers using the Recovery Self-Assessment scale | baseline, 12 months, 24 months
  This is a 32-item, self-administered rating scale that will measure perceptions about recovery principles and overall quality of services. Each item is rated on a five-point scale from 1=Strongly disagree to 5=Strongly agree. Higher scores indicate greater quality care.

SECONDARY OUTCOMES:
Change on Patient-centeredness | baseline, 12 months, 24 months
  Measured by Youth Services Survey (YSS). Each item is rated on a five-point scale from 1=Strongly disagree to 5=Strongly agree. Higher scores mean more Patient-centeredness.
Change on Medication adherence | baseline, 12 months, 24 months
  Measured by the Brief Adherence Rating Scale (BARS). It consists of 4 items: 3 questions and an overall visual analog rating scale to assess the percentage of antipsychotic medication doses taken by the user in the past month (0%-100%).
Change on Retention | baseline, 12 months, 24 months
  Measured by the Service Utilization and Resources Form (SURF). Time remaining in treatment will be estimated by counting the number of days between randomization to the time of the last mental health service received measured by the SURF. Range: from 0 to 365 days over a 12 month period; from 0 to 730 days over a 24-month period.
Change on Psychotic symptoms | baseline, 12 months, 24 months
  Measured by Positive and Negative Syndrome Scale (PANSS). This scale will be used to assess positive and negative symptoms (only the first 14 items). The level of psychopathology is rated on a seven-point scale from 1=Absent to 7=Extreme. Higher scores mean worse symptomatology.
Change on Social and Occupational Functioning | baseline, 12 months, 24 months
  Measured by the Social and Role Functioning in Psychosis and Schizophrenia (SRFP) scale. This scale asks for social, behavioral, and occupational difficulties associated with mental illness, including psychosis and schizophrenia. Functioning is rated on an eleven-point scale from 0=Extreme role dysfunction to 10=Superior social/interpersonal functioning. Higher scores mean better social and occupational functioning.
Change on Recovery Orientation | baseline, 12 months, 24 months
  Measured by the Questionnaire about the Process of Recovery (QPR). This instrument has 15 items each scored on a four-point scale ranging from 0=Strongly disagree to 4=Strongly agree. A Higher scores indicate greater recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Alvarado, MD PhD, Principal Investigator — University of Chile
Locations (1):
- CESAM San Joaquín, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
We aim to produce and share a high-quality, well-documented, and de-identified final dataset with other researchers after publication of results bearing on the specific aims of our proposal. By "high quality," we refer to our commitment to follow the guidelines on rigor and transparency by NIH to ensure strict application of the scientific method and that every effort will be made to collect data that is reliable, valid, and representative of the population studied. By "well-documented," we mean that an accessible code book will define individual variables and any scales derived from those variables, sampling plans and sampling results, procedures for handling missing data, and all other information required to use the data and to report the results with fidelity.
  By "de-identified," we mean that the data will not allow for the identification of the specific individuals who participated in this research.
Time Frame: According to NIMH guidelines.
Access Criteria: Requests for data will be directed to the study Steering Committee. We will work in consultation with the NIH staff, as well as our Steering Committee and DCC, to ensure that our data sharing protocols are in line with NIH policies on the timely release and sharing of data.

REFERENCES:
- [Derived] Mascayano F, Bello I, Andrews H, Arancibia D, Arratia T, Burrone MS, Conover S, Fader K, Jorquera MJ, Gomez M, Malverde S, Martinez-Ales G, Ramirez J, Reginatto G, Restrepo-Henao A, Rosencheck RA, Schilling S, Smith TE, Soto-Brandt G, Tapia E, Tapia T, Velasco P, Wall MM, Yang LH, Cabassa LJ, Susser E, Dixon L, Alvarado R. OnTrack Chile for people with early psychosis: a study protocol for a Hybrid Type 1 trial. Trials. 2022 Sep 5;23(1):751. doi: 10.1186/s13063-022-06661-7. PMID 36064643